CLINICAL TRIAL: NCT06397963
Title: A Single-arm Clinical Study of Autologous Tumor-Infiltrating Lymphocyte (GT307 Injection ) for Treatment of Patients With Solid Tumours
Brief Title: Autologous Tumor-Infiltrating Lymphocyte (GT307 Injection ) for Treatment of Patients With Solid Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other); Beijing GoBroad Hospital (Other); Beijing Arion Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-307-002
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT307 injection treatment group (Experimental)
  Interventions: Biological: GT307 injection

INTERVENTIONS:
Biological: GT307 injection — GT307 injection to treat solid tumours

SUMMARY:
This study is a single arm, open design aimed at evaluating the safety and tolerability of Autologous Tumor-Infiltrating Lymphocyte (GT307 injection ) for treatment of patients with solid tumours,while evaluating pharmacokinetic characteristics and efficacy assessment to determine the optimal biological dose (OBD).

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in the study, sign the informed consent form, and be willing and able to comply with the study protocol.
* 2. Aged 18-70 years old (eligibility for subjects over 70 years old shall be jointly determined by the investigator and the medical monitor of the collaborating party).
* 3. Diagnosed as patients with advanced solid tumors who have failed standard treatment, have no available standard treatment, or are unable to receive standard treatment.
* 4. Having at least one lesion that is untreated with radiotherapy or other local therapies, with accessible tumor tissue (assessed by the investigator), and from which a tissue block of ≥1.0 cm³ can be isolated after resection (either from a single lesion or a combination of multiple lesions) for the preparation of autologous tumor-infiltrating lymphocytes (TILs); minimally invasive procedures should be used whenever possible.
* 5. After tumor sampling, having at least one measurable lesion as defined by the RECIST v1.1 criteria, and the lesion must not have received radiotherapy or other local therapies (unless such therapies were administered more than 3 months prior and the lesion has demonstrated progression).
* 6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* 7. Expected survival time of ≥12 weeks.
* 8. Adequate function of major organs meeting the following requirements:

  1. Hematological parameters: Since the normal reference ranges may vary among different central laboratories, the final assessment shall be made by the investigator based on comprehensive judgment, with the following references:

     * Absolute Neutrophil Count (ANC) ≥1.0×10⁹/L;
     * Lymphocyte Count (LC) ≥0.5×10⁹/L;
     * Platelet Count (PLT) ≥80×10⁹/L;
     * Hemoglobin (Hb) ≥90 g/L.
  2. Liver function parameters: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase (ALP) ≤2.5×Upper Limit of Normal (ULN); Total Bilirubin (TBIL) ≤1.5×ULN. The criteria may be relaxed under the following circumstances:

     * For subjects with confirmed liver metastases: AST and/or ALT ≤5×ULN;
     * For subjects with confirmed liver or bone metastases: ALP ≤5×ULN;
     * For subjects with confirmed Gilbert's syndrome: TBIL ≤3.0 mg/dL.
  3. Renal function parameters: Creatinine Clearance Rate (CrCL) ≥45 mL/min (calculated using the Cockcroft-Gault formula), or serum creatinine within the normal range; and urine protein <2+.
  4. Coagulation function parameters: Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN, and International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5×ULN simultaneously.
  5. Adequate cardiac function.
  6. Adequate pulmonary function.
* 9. Non-surgically sterilized women of childbearing potential must agree to use at least one medically approved contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period and for 1 year after the end of study treatment; the serum human chorionic gonadotropin (HCG) test result of such subjects must be negative within 7 days prior to cell infusion.
* 10. Adverse reactions caused by prior treatments must have resolved to CTCAE 5.0 Grade ≤1 before tumor sampling, or be judged by the investigator and the collaborating medical team as having no interference with the study.
* 11. For subjects enrolled in the study due to disease progression, imaging documentation confirming disease progression after the last prior treatment must be available before tumor sampling.

Exclusion Criteria:

-1. Subjects with spinal cord compression that cannot be relieved by surgery and/or radiotherapy are not eligible for enrollment.

(For treated subjects, enrollment is permitted if clinical evidence demonstrates that symptoms have been relieved for ≥1 week prior to surgical sampling.)

* 2. Subjects with uncontrolled tumor-related pain as assessed by the investigator. Subjects requiring analgesic treatment must be on a stable analgesic regimen at the time of study entry. Symptomatic lesions suitable for palliative radiotherapy must be treated before study entry.
* 3. A history of bleeding events occurring within 3 months prior to screening, including but not limited to gastrointestinal bleeding caused by fundic or esophageal varices, increased bleeding risk due to portal hypertension, active gastrointestinal bleeding, etc.; or subjects assessed by the investigator as having a high risk of major bleeding (examples include but are not limited to tumors encasing or invading major blood vessels [i.e., carotid artery, jugular vein, bronchial artery] and/or exhibiting other high-risk features such as fistulas, significant cavitary lesions, a history of prior bleeding [≤60 days from signing the ICF]).
* 4. A history of arterial/venous thrombotic events occurring within 3 months prior to screening, including but not limited to cerebrovascular accident, deep vein thrombosis, and pulmonary embolism, etc.
* 5. A diagnosis of interstitial pneumonia, clinically significant active pneumonia at screening, or other respiratory system diseases that severely impair pulmonary function.
* 6. A history of clinically significant cardiovascular diseases, including but not limited to:

  1. Congestive heart failure (NYHA classification > Class 2);
  2. Unstable angina pectoris;
  3. Myocardial infarction occurring within the past 3 months;
  4. Any supraventricular or ventricular arrhythmias requiring treatment or intervention.
* 7. Subjects with ≥3 untreated central nervous system (CNS) metastases at screening.

(Enrollment is permitted if subjects have ≤3 CNS metastases, with the largest diameter <1 cm, no peritumoral edema on brain imaging (MRI or CT), and no evidence of progressive CNS disease on brain imaging for at least 3 months after treatment.)

* 8. A history of autoimmune diseases, or active autoimmune diseases requiring treatment with systemic corticosteroids or immunosuppressive agents (>10 mg/day of prednisone or equivalent).
* 9. Presence of refractory or intractable epilepsy, massive pleural effusion, ascites, pericardial effusion uncontrolled by medication, active gastrointestinal bleeding, or contraindications to IL-2 administration.
* 10. A history of malignant tumors other than the target indication within 5 years prior to screening (excluding adequately treated basal cell or squamous cell skin cancer, surgically resected ductal carcinoma in situ of the breast, etc.), unless the investigator determines that the potential benefits to the subject outweigh the risks.
* 11. A history of infectious diseases within 1 year prior to screening, such as HIV, syphilis, active viral hepatitis, active tuberculosis, active EBV and/or CMV infection; or a history of active tuberculosis infection for more than 1 year without standard treatment. Subjects with active hepatitis B or C are excluded.

HBsAg- or HBcAb-positive subjects may participate in the study if their HBV DNA test result is below the lower limit of normal (LLN) of the testing laboratory at the study site.

HCV antibody-positive subjects may participate if their HCV RNA test result is below the LLN of the testing laboratory at the study site.

For carriers enrolled in the study, antiviral treatment should be arranged as appropriate, and regular nucleic acid copy number quantitative testing should be performed during the study period.

* 12. Subjects with a history of prior allogeneic bone marrow transplantation or solid organ transplantation.
* 13. Use of anti-angiogenic agents (e.g., bevacizumab, a VEGF inhibitor) within 4 weeks prior to sampling.
* 14. Receipt of systemic anti-tumor therapy within 4 weeks prior to lymphodepletion conditioning, except for the following circumstances:

  * Bridge therapy;
  * If prior treatment included nitrosourea or mitomycin chemotherapy, the interval between the end of chemotherapy and the expected first study treatment administration must be at least 6 weeks for enrollment;
  * If prior treatment included small-molecule targeted therapy, the interval between the end of treatment and the expected first study treatment administration must be at least 5 half-lives of the drug for enrollment.
* 15. Prior receipt of genetically modified or edited cell therapy products (excluding autologous immune cell therapy products without genetic modification or editing that were administered more than 1 year before the date of cell infusion).
* 16. A history of hypersensitivity reactions to any component of the drugs intended for use in the study, including but not limited to autologous tumor-infiltrating lymphocytes (TILs), cyclophosphamide, fludarabine, interleukin-2 (IL-2), dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40, and antibiotics (β-lactam antibiotics, gentamicin).
* 17. A known history of mental illness, alcoholism, drug addiction, or substance abuse, etc.
* 18. A history of grade 3 or higher adverse reactions from prior immunotherapy that failed to resolve to CTCAE Grade 1 or lower within 28 days; any disease or condition (including other illnesses, metabolic disorders, physical examination findings, or abnormal laboratory test results) that would reasonably raise suspicion of contraindicating the use of study drugs, interfere with the interpretation of study results, or place the subject at high risk of treatment-related complications.
* 19. Pregnant or lactating women; or women planning to become pregnant, lactate, or conceive within 1 year after cell infusion.
* 20. Receipt of other investigational drugs/study treatments within 4 weeks prior to screening, or plans to participate in other investigational drugs/study treatments during the study period.
* 21. Other circumstances deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-04-18 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adcersed events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection（GT307) in patients with relapsed/metastatic advanced solid tumor as measured by the incidence and severity of adcersed events per CTCAE 5.0

SECONDARY OUTCOMES:
Objective response rate | 3 years
  To evaluate efficacy parameters such Objective Response Rate (ORR) per RECIST 1.1, as assessed by the Investigator

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Arion Cancer Center, Beijing, Beijing Municipality
  - Beijing GoBroad hospital, Beijing, Beijing Municipality
  - The Affiliated Hospital Of Xuzhou Medical University, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No